CLINICAL TRIAL: NCT04023955
Title: Feasibility of a Twitter Campaign to Promote HPV Vaccine Uptake Among Racially/Ethnically Diverse Young Adult Women Living in Public Housing
Brief Title: Promoting HPV Vaccine Through Twitter
Status: Completed | Type: Observational
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Jennifer Allen, Professor, Tufts University
Other Study IDs: 1603045
Record Dates: First submitted 2019-07-01; First posted 2019-07-18 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Human Papilloma Virus
Keywords: vaccination; feasibility; public housing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention: Twitter messages delivered over 1 month period
  Interventions: Behavioral: Twitter

INTERVENTIONS:
Behavioral: Twitter — Participants received a daily tweet over a period of one-month with educational messages about HPV vaccine and cervical cancer

SUMMARY:
This study assessed the feasibility of implementing a one-month Twitter campaign to promote knowledge about the human papillomavirus (HPV) vaccine among low-income women living in public housing.

DETAILED DESCRIPTION:
Investigators recruited a convenience sample (n=35) of women ages 18-26 years who resided in public housing in Massachusetts. Investigators assessed the feasibility and acceptability of the campaign. Online assessed changes in HPV knowledge, attitudes, and vaccine intentions before and after the campaign.

ELIGIBILITY:
Inclusion Criteria:

English-speaking women Age18-26 years Residents of public housing in two Massachusetts cities

Ages: 18 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Women residing in public housing Ages18-26 years No history of cervical cancer
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-06-10 (Actual); Study Completion 2018-06-10 (Actual)

PRIMARY OUTCOMES:
Measure of Humanpapilloma VirusVaccine Knowledge | 3 months
  13 items that assess knowledge about HPV, the HPV vaccine, and cervical cancer; HPV and cervical cancer risk factors and HPV transmission. Score from 0-100% with higher scores indicating greater knowledge

IPD SHARING:
Plan to Share IPD: No